CLINICAL TRIAL: NCT07218094
Title: Neuromechanical Mechanisms of Exosuit-assisted Gait Rehabilitation After Stroke
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Lou Awad, PT, DPT, PhD, Associate Professor, Boston University Charles River Campus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4440
Record Dates: First submitted 2025-10-02; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Stroke
Keywords: Stroke; Gait Disorders, Neurologic; Gait Analysis; Neuromuscular Control; Rehabilitation, Stroke; Exoskeleton Device; Biomechanics
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Participants will complete a 3-minute treadmill walking trial without robotic exosuit assistance and then complete two trials with different assistance profiles from which a preferred profile will be identified.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Walking without robotic ankle assistance (Active Comparator): Subjects will complete a 3-minute treadmill walking trial without any intervention
  Interventions: Device: Walking with robotic ankle assistance

INTERVENTIONS:
Device: Walking with robotic ankle assistance — Subjects will complete two trials of 3-minute treadmill walking with active robotic exosuit assistance, from which a preferred assistance profile will be identified. The treadmill walk associated with the preferred profile will be used for primary analyses.

SUMMARY:
Stroke survivors often experience impaired neuromechanical control that limits walking speed and quality, particularly due to deficits in paretic propulsion. This study aims to identify patient-specific neuromechanical locomotor control strategies, link them to biomechanical gait impairments, and investigate how these strategies influence responses to soft robotic exosuit assistance of paretic propulsion and ground clearance during walking. The study focuses on adults who are more than six months post-stroke and have observable gait deficits.

The main questions are:

1. How do neuromechanical control patterns (i.e., electromyography-measured muscle coordination) affect walking speed, quality, and gait biomechanics after stroke?
2. Do individuals with distinct neuromechanical patterns respond differently to robotic exosuit-assisted gait rehabilitation?

Researchers will compare walking performance without and with robotic exosuit assistance to determine whether tailoring exosuit-assisted gait intervention to patient-specific neuromechanical profiles can lead to greater improvements in walking function. Participants will complete treadmill and overground walking assessments instrumented with motion capture, EMG, and force plates, performing one trial without assistance and two trials with robotic exosuit assistance delivered at different assistance onset timings, from which a preferred assistance setting will be identified. The walking trial associated with the preferred assistance setting will be used for primary analyses.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* >6 months post-stroke
* Observable gait deficits
* Able to walk overground and on a treadmill without body-weight support
* Able to communicate clearly with investigators and follow instructions
* Able to fit the exosuit components, including height between 4'8" and 6'7", weight < 264lbs, neutral ankle dorsiflexion during standing.

Exclusion Criteria:

* Comorbidities besides stroke that impair walking (musculoskeletal, cardiovascular, pulmonary, or neurological)
* Severe pain, neglect, hemianopia, or aphasia limiting comprehension
* Unexplained dizziness or more than 2 falls in the previous month
* Inability to communicate (as assessed by a licensed physical therapist)
* Inability to wear the exosuit due to conditions that require medical management, such as open wounds or broken skin, or as assessed by a licensed physical therapist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dynamic Motor Control Index (DMCI) | Assisted - Baseline
  Difference in neuromuscular control quality compared to normative data with and without exosuit
Correlation Between Propulsion and Weight-Acceptance Motor Modules (Temporal) | Assisted - Baseline
  Difference in the merging of motor module structures quantified by correlation coefficient between the propulsion temporal module and weight-acceptance temporal module, computed from EMG data by non-negative matrix factorization, with and without exosuit
Correlation Between Weight-Acceptance and Swing-Limb Deceleration Motor Modules (Temporal) | Assisted - Baseline
  Difference in the merging of motor module structures quantified by correlation coefficient between the weight-acceptance temporal module and swing-limb deceleration temporal module, computed from EMG data by non-negative matrix factorization, with and without exosuit
Variance Accounted For (VAF) by Four Muscle Synergies | Assisted - Baseline
  Difference in the variance in muscle activation accounted for by the 4-synergy model, measuring the quantitative shift in muscle coordination complexity with and without exosuit (%)
Paretic Propulsion | Assisted - Baseline
  Difference in anterior-posterior ground reaction force with and without exosuit (N)

SECONDARY OUTCOMES:
Joint Angle | Assisted - Baseline
  Difference in joint angles computed using inverse dynamics, including ankle, knee, and hip angles, with and without exosuit (degrees)
Joint Torque | Assisted - Baseline
  Difference in joint torques computed using inverse dynamics, including ankle, knee, and hip torques, with and without exosuit (Nm/kg)
Joint Power | Assisted - Baseline
  Difference in joint power computed using inverse dynamics, including ankle, knee, and hip power, with and without exosuit (W/kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Boston University Neuromotor Recovery Laboratory, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified subject data with and without robotic ankle exosuit assistance may be published as part of the manuscript. Data may include kinematics, kinetics, and clinical data.
Time Frame: At the time of manuscript acceptance

REFERENCES:
- [Background] Awad LN, Esquenazi A, Francisco GE, Nolan KJ, Jayaraman A. The ReWalk ReStore soft robotic exosuit: a multi-site clinical trial of the safety, reliability, and feasibility of exosuit-augmented post-stroke gait rehabilitation. J Neuroeng Rehabil. 2020 Jun 18;17(1):80. doi: 10.1186/s12984-020-00702-5. PMID 32552775
- [Background] Farris DJ, Hampton A, Lewek MD, Sawicki GS. Revisiting the mechanics and energetics of walking in individuals with chronic hemiparesis following stroke: from individual limbs to lower limb joints. J Neuroeng Rehabil. 2015 Feb 27;12:24. doi: 10.1186/s12984-015-0012-x. PMID 25889030
- [Background] Hsiao H, Awad LN, Palmer JA, Higginson JS, Binder-Macleod SA. Contribution of Paretic and Nonparetic Limb Peak Propulsive Forces to Changes in Walking Speed in Individuals Poststroke. Neurorehabil Neural Repair. 2016 Sep;30(8):743-52. doi: 10.1177/1545968315624780. Epub 2015 Dec 31. PMID 26721869
- [Background] Bowden MG, Balasubramanian CK, Neptune RR, Kautz SA. Anterior-posterior ground reaction forces as a measure of paretic leg contribution in hemiparetic walking. Stroke. 2006 Mar;37(3):872-6. doi: 10.1161/01.STR.0000204063.75779.8d. Epub 2006 Feb 2. PMID 16456121
- [Background] Porciuncula F, Arumukhom Revi D, Baker TC, Sloutsky R, Walsh CJ, Ellis TD, Awad LN. Effects of high-intensity gait training with and without soft robotic exosuits in people post-stroke: a development-of-concept pilot crossover trial. J Neuroeng Rehabil. 2023 Nov 7;20(1):148. doi: 10.1186/s12984-023-01267-9. PMID 37936135
- [Background] Awad LN, Kudzia P, Revi DA, Ellis TD, Walsh CJ. Walking faster and farther with a soft robotic exosuit: Implications for post-stroke gait assistance and rehabilitation. IEEE Open J Eng Med Biol. 2020;1:108-115. doi: 10.1109/ojemb.2020.2984429. Epub 2020 Apr 2. PMID 33748765
- [Background] Moucheboeuf G, Griffier R, Gasq D, Glize B, Bouyer L, Dehail P, Cassoudesalle H. Effects of robotic gait training after stroke: A meta-analysis. Ann Phys Rehabil Med. 2020 Nov;63(6):518-534. doi: 10.1016/j.rehab.2020.02.008. Epub 2020 Mar 27. PMID 32229177
- [Background] Collimore AN, Aiello AJ, Pohlig RT, Awad LN. The Dynamic Motor Control Index as a Marker of Age-Related Neuromuscular Impairment. Front Aging Neurosci. 2021 Jul 22;13:678525. doi: 10.3389/fnagi.2021.678525. eCollection 2021. PMID 34366824
- [Background] Steele KM, Rozumalski A, Schwartz MH. Muscle synergies and complexity of neuromuscular control during gait in cerebral palsy. Dev Med Child Neurol. 2015 Dec;57(12):1176-82. doi: 10.1111/dmcn.12826. Epub 2015 Jun 17. PMID 26084733
- [Background] Bizzi E, Cheung VC. The neural origin of muscle synergies. Front Comput Neurosci. 2013 Apr 29;7:51. doi: 10.3389/fncom.2013.00051. eCollection 2013. PMID 23641212
- [Background] Allen JL, Kautz SA, Neptune RR. The influence of merged muscle excitation modules on post-stroke hemiparetic walking performance. Clin Biomech (Bristol). 2013 Jul;28(6):697-704. doi: 10.1016/j.clinbiomech.2013.06.003. Epub 2013 Jul 2. PMID 23830138
- [Background] Neptune RR, Clark DJ, Kautz SA. Modular control of human walking: a simulation study. J Biomech. 2009 Jun 19;42(9):1282-7. doi: 10.1016/j.jbiomech.2009.03.009. Epub 2009 Apr 25. PMID 19394023
- [Background] Ting LH, Chiel HJ, Trumbower RD, Allen JL, McKay JL, Hackney ME, Kesar TM. Neuromechanical principles underlying movement modularity and their implications for rehabilitation. Neuron. 2015 Apr 8;86(1):38-54. doi: 10.1016/j.neuron.2015.02.042. PMID 25856485
- [Background] Sloot LH, Baker LM, Bae J, Porciuncula F, Clement BF, Siviy C, Nuckols RW, Baker T, Sloutsky R, Choe DK, O'Donnell K, Ellis TD, Awad LN, Walsh CJ. Effects of a soft robotic exosuit on the quality and speed of overground walking depends on walking ability after stroke. J Neuroeng Rehabil. 2023 Sep 1;20(1):113. doi: 10.1186/s12984-023-01231-7. PMID 37658408
- [Background] Awad LN, Lewek MD, Kesar TM, Franz JR, Bowden MG. These legs were made for propulsion: advancing the diagnosis and treatment of post-stroke propulsion deficits. J Neuroeng Rehabil. 2020 Oct 21;17(1):139. doi: 10.1186/s12984-020-00747-6. PMID 33087137
- [Background] Allen JL, Kautz SA, Neptune RR. Step length asymmetry is representative of compensatory mechanisms used in post-stroke hemiparetic walking. Gait Posture. 2011 Apr;33(4):538-43. doi: 10.1016/j.gaitpost.2011.01.004. Epub 2011 Feb 11. PMID 21316240
- [Background] Moore SA, Boyne P, Fulk G, Verheyden G, Fini NA. Walk the Talk: Current Evidence for Walking Recovery After Stroke, Future Pathways and a Mission for Research and Clinical Practice. Stroke. 2022 Nov;53(11):3494-3505. doi: 10.1161/STROKEAHA.122.038956. Epub 2022 Sep 7. PMID 36069185
- [Background] Kesar T. The Effects of Stroke and Stroke Gait Rehabilitation on Behavioral and Neurophysiological Outcomes:: Challenges and Opportunities for Future Research. Dela J Public Health. 2023 Aug 31;9(3):76-81. doi: 10.32481/djph.2023.08.013. eCollection 2023 Aug. PMID 37701480
- [Background] Clark DJ, Ting LH, Zajac FE, Neptune RR, Kautz SA. Merging of healthy motor modules predicts reduced locomotor performance and muscle coordination complexity post-stroke. J Neurophysiol. 2010 Feb;103(2):844-57. doi: 10.1152/jn.00825.2009. Epub 2009 Dec 9. PMID 20007501